CLINICAL TRIAL: NCT07026123
Title: A Real-world Study of Liposomal Irinotecan (Onivyde)-Based Therapy in Patients With Locally Advanced/Metastatic Pancreatic Cancer in China
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Servier (Tianjin) Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: IIT-95013-002-CHN
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Advanced Pancreatic Cancer
Keywords: Pancreatic Cancer; chemotherapy; liposomal irinotecan; real world research
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irinotecan sucrosofate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Liposomal irinotecan (Onivyde®)-based treatment.
  Interventions: Drug: Nal-IRI (Onivyde®)-based treatment
- Control group: Real medication data from accepting other second-line treatment options in the China Pancreas Data Center (CPDC) project.
  Interventions: Drug: Other second-line treatment

INTERVENTIONS:
Drug: Nal-IRI (Onivyde®)-based treatment — Nal-IRI (Onivyde®) combined with 5-FU/LV is used for metastatic pancreatic ductal adenocarcinoma patients who have progressed after treatment with gemcitabine. The recommended dose of Nal-IRI (Onivyde®) is 70 mg/m^2, administered intravenously for 90 minutes, once every 2 weeks. In patients known to be homozygous for the UGT1A1 * 28 allele, the recommended starting dose of Nal-IRI (Onivyde®) is 50 mg/m^2, administered intravenously within 90 minutes. Based on tolerance, increase the dose of Nal-IRI (Onivyde®) to 70 mg/m^2 in subsequent cycles.
  Groups: Experimental group
Drug: Other second-line treatment — Other second-line treatment
  Groups: Control group

SUMMARY:
This study is designed to evaluate the real world efficacy and safety of the liposomal irinotecan (Onivyde®)-based treatment scheme in Chinese patients with locally advanced or metastatic pancreatic cancer, and to compare the efficacy with that of the whole pancreatic cancer population who did not receive relevant treatment.

DETAILED DESCRIPTION:
Chinese patients with pancreatic cancer are mostly treated according to foreign clinical research, lacking the diagnosis and treatment data of efficacy and safety of Chinese population. In the NAPOLI-1 study, irinotecan liposomes (Onivyde®) The combination of 5-fluorouracil and folinic acid (Nal-IRI+5-FU/LV) has shown survival benefits in patients with metastatic pancreatic ductal adenocarcinoma (mPDAC) who have previously received gemcitabine-based treatment. The NAPOLI-3 study showed that NALIRIFOX (Nal-IRI+oxaliplatin+5-FU/LV) significantly improved overall survival (OS) and progression free survival (PFS) compared to albumin bound paclitaxel and gemcitabine in newly diagnosed mPDAC patients. However, the efficacy and safety data of Nal-IRI-based treatment regimens in China are limited. In August 2023, Onivyde® was commercially listed in China. The purpose of this study is to: ① evaluate the real world efficacy and safety of Onivyde®-based treatment schemes in Chinese patients with locally advanced or metastatic pancreatic cancer; ② analyze the efficacy of Onivyde® treatment and the efficacy of all pancreatic cancer patients who have not received relevant treatment using the project data of China Advanced pancreatic cancer Big Data Center (Renji Hospital Cancer Department is the national leading unit), in conjunction with the survival follow-up data of China Center for Disease Control and Prevention of Chronic Non communicable Diseases.

ELIGIBILITY:
Inclusion Criteria of the experimental group:

* Age ≥ 18 years old.
* Patients with locally advanced or metastatic PDAC diagnosed by pathology.
* Patients who received at least one cycle of Nal-IRI (Onivyde®）+ 5-FU/LV treatment.
* Patients who have progressed in treatment with gemcitabine or gemcitabine containing regimens in the past.
* The patient voluntarily participates in the study and signs an informed consent form.

Inclusion Criteria of the control group:

* Age ≥ 18 years old.
* Patients with locally advanced or metastatic PDAC diagnosed by pathology.
* Not received Nal IRI (Onivyde®)+ 5-FU/LV treatment in the past.

Exclusion Criteria:

* Confirm pregnant or lactating women.
* The patient's clinical data is not available.
* The researchers determined that they were not suitable for inclusion in the study due to other circumstances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Experimental group: 40 patients Control group: Depends on the real world condition of China Pancreas Data Center (CPDC) project.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 24 months
  Overall Survival (OS) is defined as the time from enrollment to death from any cause.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 24 months
  Progression-Free Survival (PFS) is defined as the time from first-dose to the first documented disease progression or death
Time To Progress (TTP) | Up to 24 months
  Time To Progress (TTP) is defined as the length of time from first-dose until the date of disease progression
Overall Response Rate (ORR) | Up to 24 months
  Overall Response Rate (ORR) is defined as the percentage of people in this study who have a partial response or complete response (according to RESIST v1.1) to the treatment
Disease Control Rate (DCR) | Up to 24 months
  Disease Control Rate (DCR) is defined as the proportion of patients with complete response, partial response or stable disease, according to RESIST v1.1
Safety and tolerability by incidence, severity and outcome of adverse events | Until 30 day safety follow-up visit
  Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Liwei Wang, M.D., Principal Investigator — Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No